CLINICAL TRIAL: NCT03206619
Title: Study on Patient Acceptance and Engagement of Timely Tailored Motivational Messages Sent by a Health Recommender System and Delivered Via a Mobile App for Smoking Cessation
Brief Title: A Health Recommeder System to Tailor Message Preferences in a Smoking Cessation Programme
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); Salumedia Tecnologías (Unknown); Aristotle University Of Thessaloniki (Other); Northern Greece Neurofeedback Center (Unknown)
Responsible Party: Principal Investigator, Santiago Hors-Fraile, Principal Investigator, University of Seville
Other Study IDs: H2020-681120
Record Dates: First submitted 2017-02-07; First posted 2017-07-02 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Smoking Cessation; Health Behavior; Smoking, Tobacco; Smoking
Keywords: smoking; habit; preference; behavior; tailoring; cessation; engagement; digital; mobile app; recommender system
MeSH Terms: conditions — Smoking Cessation; Health Behavior; Tobacco Smoking; Smoking; Habits; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Social, Local and Mobile: Patients having smoking cessation standard care (behavioral and pharmacological therapy) and using the SoLoMo mobile app that sends them motivational messages.
  Interventions: Other: Social, Local and Mobile

INTERVENTIONS:
Other: Social, Local and Mobile — Patients in a smoking cessation program will use a mobile application to receive messages and rate them from their smartphones. The messages patient will receive belong to one of the following five topics: general motivation, diet tips, physical exercise tips, personal performance, and the benefits of being a non-smoker. For each one of these topics, there will be a pool of 150 different messages with tailored information for the patient. Topics and messages were approved by a smoking cessation psychologist and a pulmonologist. The selection of the time the messages have to be sent, and the message topic is selected by an health recommender system algorithm based on the patients' user profile (demographic information, message rating information, and app interaction information).
  Other Names: SoLoMo

SUMMARY:
Patients attending the smoking cessation programme at the Virgen del Rocío University Hospital under the SoLoMo clinical trial of the SmokeFreeBrain project and provided with the SoLoMo mobile app will be observed for one year. This mobile app which sends the patients tailored health motivational messages selected by a health recommender system, and based on their user profile retrieved from an electronic health record. Patients' messages feedback and interactions with the app will be analyzed and evaluated following an observational prospective methodology to see whether patients like the messages, and measure the patient engagement with the health recommender system.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be taken from the the smoking cessation unit of the Virgen del Rocio University Hospital (Seville, Spain)
* Patients must be willing to start the treatment to quit smoking
* Patients must own an Android smartphone and be able to interact with it
* Patients must be willing to and install the "Libre de Humos" smoking cessation app recommended by the doctor in the SmokeFreeBrain study.
* Patients must sign an informed consent

Exclusion Criteria:

* Patients have known previous adverse effects on the pharmacological treatment included in the study (Bupropion & Varenicline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult smokers living in Seville (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Objective quality of the health recommender system | Up to 18 months
  The objective quality of the health recommender system is calculated by measuring its precision. The precision of the health recommender system is the relation between the number of messages patients have rated with positive and/or positive and neutral feedback the first month (baseline), and all subsequent months.
Subjective quality of the health recommender system | Up to 18 months
  The subjective quality of the health recommender systems is determined by eighteen questions which will be answered using a 1 to 5 point Likert scale by all patients finishing their smoking cessation programme.
Engagement at aggregated level - Mobile application rolling retention | Up to 18 months
  The percentage of users still active N days after installation. This is a ratio of the number of users whose last day of activity is past day N to the number of users who could have been active on day N. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application session length distribution | Up to 18 months
  The session length is defined as the length of time between the start of the application event and the end of the application event. The session length determines the engagement as it is relevant to know how much time patients spend in the app per session. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Mobile application usage frequency | Up to 18 months
  The frequency of use is a measure of how often each unique patient used the app within a given time interval. This metric will be assessed throughout the observation until its end.
Engagement at aggregated level - Number of sessions per user | Up to 18 months
  A session is one use of the mobile application by a patient. This begins when the application is launched and ends when the application is terminated. This metric will be assessed throughout the observation
  until its end.
Engagement at aggregated level - Return rate | Up to 18 months
  Return rate measures the percentage of patients who return to the app on a specific time after installation. It is measured by cohort group - that is, based on when patients first opened the app. It is calculated as the ratio of the number of users active on a given period to the size of the cohort. This metric will be assessed throughout the observation until its end.
Engagement at individual level | Up to 18 months
  Engagement at individual level will be assessed based on the rate of read messages by the patients. This is calculated as the quotient between the messages the patients have read, and the total number of messages the system has sent to the patients. This metric will be assessed throughout the observation until its end.

CONTACTS AND LOCATIONS:
Locations (1):
- Virgen del Rocío University Hospital, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
An anonymized subset of the database will be made available 5 years after the completion of the project. This embargo period aims to support a correct IPR management within the SmokeFreeBrain consortium, as well as to guarantee the availability of the dataset to the SmokeFreeBrain researchers in order to leverage the scientific production related to the project outcomes. The database can be shared at the end of the embargo period but specific consent will be required. The informed consent form and the information sheet provided to the participants will inform them regarding this attribute of the data.

REFERENCES:
- [Derived] Hors-Fraile S, Schneider F, Fernandez-Luque L, Luna-Perejon F, Civit A, Spachos D, Bamidis P, de Vries H. Tailoring motivational health messages for smoking cessation using an mHealth recommender system integrated with an electronic health record: a study protocol. BMC Public Health. 2018 Jun 5;18(1):698. doi: 10.1186/s12889-018-5612-5. PMID 29871595
- See also: Official website of the original project — http://www.smokefreebrain.eu